CLINICAL TRIAL: NCT06109038
Title: Effects of ITB Myofascial Release on Symptoms Associated With Knee OA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nida Anwar / REC-01686
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee OA; ITB tightness; Graston technique
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- : Conventional PT + ITB release with graston technique (Experimental): An emollient will be applied to the leg from the lateral joint line along the tibial condyle to just below the iliac crest. The instrument GT-4 will be used for treatment. The tool was used to assess the soft tissue in three locations on the lateral leg: anterior to the ITB, over the ITB, and posterior to the ITB. Brushing and strumming strokes were performed to the tissue utilising the instrument's convex surface. Treatment time with the instrument is 8 -10 mins .
  Conventional PT including Hot Pack for 5mins. Quadriceps setting exercises, short arc terminal knee extension, straight leg raise, ROM excercises, hamstring curls in prone lying position, quadriceps strengthening in high sitting position, gastrocnemius muscle stretching (10reps × 5sec × 2sets). Maitland mobilization (Grade 1, 2 and 3 for 10 repititions).
  Interventions: Other: Conventional PT + ITB release with graston technique
- Conventional PT (Other): Conventional PT including Hot Pack for 5mins. Quadriceps setting exercises, short arc terminal knee extension, straight leg raise, ROM excercises, hamstring curls in prone lying position, quadriceps strengthening in high sitting position, gastrocnemius muscle stretching (10reps × 5sec × 2sets). Maitland mobilization (Grade 1, 2 and 3 for 10 repititions).
  Interventions: Other: Conventional PT

INTERVENTIONS:
Other: Conventional PT + ITB release with graston technique — An emollient will be applied to the leg from the lateral joint line along the tibial condyle to just below the iliac crest. The instrument GT-4 will be used for treatment. The tool was used to assess the soft tissue in three locations on the lateral leg: anterior to the ITB, over the ITB, and posterior to the ITB. Brushing and strumming strokes were performed to the tissue utilising the instrument's convex surface. Treatment time with the instrument is 8 -10 mins .
  Conventional PT including Hot Pack for 5mins. Quadriceps setting exercises, short arc terminal knee extension, straight leg raise, ROM exercises, hamstring curls in prone lying position, quadriceps strengthening in high sitting position, gastrocnemius muscle stretching (10reps × 5sec × 2sets). Maitland mobilization (Grade 1, 2 and 3 for 10 repetitions).
  Arms: : Conventional PT + ITB release with graston technique
Other: Conventional PT — Conventional PT including Hot Pack for 5mins. Quadriceps setting exercises, short arc terminal knee extension, straight leg raise, ROM exercises, hamstring curls in prone lying position, quadriceps strengthening in high sitting position, gastrocnemius muscle stretching (10reps × 5sec × 2sets). Maitland mobilization (Grade 1, 2 and 3 for 10 repetitions).
  Arms: Conventional PT

SUMMARY:
The aim of this randomized controlled trial is to determine the effects of ITB myofascial release with graston technique on symptoms associated with knee Osteoarthritis for reducing pain, enhancing knee range of motion and decrease functional disability.

DETAILED DESCRIPTION:
Graston technique, Instrument assisted soft tissue mobilization (IASTM) also known as myofascial release technique is a skilled myofascial intervention used for soft-tissue treatment. Graston is a myofascial release tool that decreases adhesions, trigger points and tension in muscles. Graston Technique on Iliotibial Band Syndrome resulted in a decrease in subjective symptoms and an improvement in muscle function.

ELIGIBILITY:
Inclusion Criteria:

* knee OA Grade 2 and Grade 3 according to kellgren and Lawrence grading scale
* Positive Ober's test

Exclusion Criteria:

* Patient with cardiovascular or medical illness.
* Patient with any severe trauma or surgery of knee.
* Knee deformity
* Low back pain with or without radiculopathy.
* Neurological illness
* Participants having any wound or scar on the site of treatment.
* Pregnant female
* Participants having co-morbidities such as neoplasm etc.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
WOMAC questionnaire | 4 WEEKS
  The WOMAC is a reliable , valid, and responsive instrument for evaluating the severity of OA of the knee, with metric properties. The WOMAC measures 5 items for pain (score range 0-20), 2 for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68),
Numeric Pain Rating Scale | 4 WEEKS
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain
Goniometer | 4 WEEKS
  It is an instrument that measures the available range of motion at a joint.

CONTACTS AND LOCATIONS:
Overall Officials: Maria khalid, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No